CLINICAL TRIAL: NCT05819086
Title: Motivating Change in Aging African American Smokers - Testing Messages
Brief Title: Message Testing in Aging African American Smokers
Acronym: MCAAAS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Centiment LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0217; SMPH/MEDICINE/GEN INT MD (Other: UW Madison); Version date 2/6/2023 (Other: UW Madison)
Record Dates: First submitted 2023-04-04; First posted 2023-04-19 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- "Big tobacco" video message and flyer (Active Comparator): Participants will view a "Big tobacco" video message and flyer.
  Interventions: Behavioral: Rate Emotional Response; Behavioral: Rate Impact of Message
- "It's never too late" video message and flyer (Active Comparator): Participants will view a "It's never too late" video message and flyer.
  Interventions: Behavioral: Rate Emotional Response; Behavioral: Rate Impact of Message
- Placebo Message (Placebo Comparator): Participants will view a water advertisement and flyer.
  Interventions: Behavioral: Rate Emotional Response; Behavioral: Rate Impact of Message
- Fear message video and flyer (Active Comparator): Participants will view a fear message video and flyer.
  Interventions: Behavioral: Rate Emotional Response; Behavioral: Rate Impact of Message

INTERVENTIONS:
Behavioral: Rate Emotional Response — Participants will view their assigned video package, and will be asked to rate their emotional response to the message
  Other Names: Video message and flyer
Behavioral: Rate Impact of Message — Participants will view their assigned video package, and will be asked to rate the impact of the presented messages on motivation to quit smoking.
  Other Names: Video message and flyer

SUMMARY:
The goal of this study is to examine different messages to motivate smokers who self-identify as an African American current smoker, between the ages of 50-80 years old to quit smoking. Participants will be asked to complete a survey and look at two messages.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker (smoking at least some days per week)
* Ability to read and write English
* Between the ages of 50 and 80 years old
* Self identify as African American.

Exclusion Criteria:

* History of Mild Cognitive Impairment or dementia

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Johnson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | "Big Tobacco" Video Message and Flyer | "It's Never Too Late" Video Message and Flyer | Placebo Message | Fear Message Video and Flyer
Started | 219 | 207 | 210 | 203
Completed | 219 | 207 | 210 | 203
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Big Tobacco" Video Message and Flyer | "It's Never Too Late" Video Message and Flyer | Placebo Message | Fear Message Video and Flyer | Total
Number analyzed (Participants) | 219 | 207 | 210 | 203 | 839
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 170 | 161 | 51 | 156 | 538
  >=65 years | 49 | 46 | 159 | 47 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.32 (6.652) | 58.91 (6.901) | 59.55 (6.778) | 59.40 (6.742) | 59.30 (6.759)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  cisgender Man | 97 | 83 | 96 | 88 | 364
  cisgender Woman | 112 | 115 | 106 | 109 | 442
  Non-binary | 2 | 2 | 1 | 1 | 6
  Other | 1 | 3 | 5 | 2 | 11
  Refused/Missing | 5 | 4 | 2 | 1 | 12
  transgender Man | 1 | 0 | 0 | 0 | 1
  transgender Woman | 1 | 0 | 0 | 2 | 3
Race/Ethnicity, Customized [Number; unit: Endorsements] — Endorsing Black/African American race was an inclusion criteria for the study. Additionally, the following question was asked: "Which racial group do you most strongly identify with **(choose all that apply)**?: White/Caucasian; Native Hawaiian/Pacific Islander; Asian; Native American/Alaska Native; other; refused.
  Endorsements
    Black or African American | 219 | 207 | 210 | 203 | 839
    White or Caucasian | 3 | 2 | 5 | 1 | 11
    Native American/Alaska Native | 3 | 3 | 4 | 4 | 14
    Asian | 0 | 0 | 0 | 0 | 2
    Native Hawaiian/Pacific Islander | 0 | 0 | 0 | 0 | 0
    Other | 0 | 1 | 0 | 0 | 1
    Refused | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 219 | 207 | 210 | 203 | 839

OUTCOME MEASURES:

1. Primary Outcome: Motivation to Quit Smoking
Description: Change in participants' motivation to quit pre- and post-viewing of the experimental flyer and video, using a 1 item scaled measurement of motivation to quit (1-7 scale, 7 indicating higher motivation) measured in a single online survey (~15 minutes).
Time Frame: data collected before and after intervention (baseline and approximately 15 minutes later)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Big Tobacco" Video Message and Flyer | "It's Never Too Late" Video Message and Flyer | Placebo Message | Fear Message Video and Flyer
Number analyzed (Participants) | 213 | 205 | 203 | 201
score on a scale | .3052 (1.3722) | .3220 (1.1605) | .3202 (1.2785) | .4378 (1.4448)

2. Primary Outcome: Emotional Response - Sad
Description: Measure participants' emotional response to the messages using a 1-9 scaled measurement of 14 different emotions (9 indicating more emotional response).
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 217 | 202 | 207
score on a scale | 1.281 (1.018) | 3.77 (2.800) | 3.27 (2.514) | 2.88 (2.419)

3. Primary Outcome: Emotional Response - Angry
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 218 | 202 | 207
score on a scale | 1.25 (.972) | 3.70 (2.810) | 2.189 (2.042) | 2.20 (2.093)

4. Primary Outcome: Emotional Response - Afraid
Description: Measure participants' emotional response to the messages using a 1-9 scaled measurement of 14 different emotions (9 indicating more emotional response). Emotionality will be presented together summarizing the mean presentation of these emotions by the different groups.
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 217 | 202 | 205
score on a scale | 1.252 (.947) | 3.548 (2.804) | 3.441 (2.614) | 3.210 (2.655)

5. Primary Outcome: Emotional Response - Guilty
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 215 | 202 | 206
score on a scale | 1.424 (1.232) | 4.019 (2.861) | 3.490 (2.617) | 3.524 (2.726)

6. Primary Outcome: Emotional Response - Disgusted
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 217 | 202 | 206
score on a scale | 1.410 (1.270) | 4.203 (2.916) | 2.465 (2.662) | 2.742 (2.441)

7. Primary Outcome: Emotional Response - Worried
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 218 | 202 | 206
score on a scale | 1.357 (1.137) | 4.431 (2.787) | 3.960 (2.673) | 3.700 (2.724)

8. Primary Outcome: Emotional Response - Ashamed
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 218 | 202 | 207
score on a scale | 1.357 (1.158) | 3.514 (2.666) | 2.777 (2.298) | 2.841 (2.541)

9. Primary Outcome: Emotional Response - Confused
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 218 | 202 | 207
score on a scale | 1.543 (1.568) | 2.037 (2.043) | 1.856 (1.703) | 1.773 (1.623)

10. Primary Outcome: Emotional Response - Amused
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 218 | 202 | 206
score on a scale | 4.362 (2.701) | 2.037 (2.043) | 2.080 (2.026) | 2.471 (2.419)

11. Primary Outcome: Emotional Response - Hopeful
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 217 | 201 | 207
score on a scale | 4.324 (2.674) | 5.189 (2.608) | 4.906 (2.588) | 5.174 (2.771)

12. Primary Outcome: Emotional Response - Motivated
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 216 | 201 | 207
score on a scale | 4.695 (2.827) | 5.380 (2.576) | 5.060 (2.696) | 5.073 (2.657)

13. Primary Outcome: Emotional Response - Understood
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 209 | 215 | 201 | 206
score on a scale | 5.024 (3.015) | 5.800 (2.637) | 5.741 (2.770) | 5.738 (2.594)

14. Primary Outcome: Emotional Response - Happy
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 209 | 216 | 200 | 205
score on a scale | 5.057 (2.597) | 2.912 (2.580) | 2.940 (2.391) | 3.102 (2.502)

15. Primary Outcome: Emotional Response - Surprised
Description: as for outcome 2
Time Frame: data collected at one time point, post-intervention, up to approximately 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Message | "Big Tobacco" Video Message and Flyer | Fear Message Video and Flyer | "It's Never Too Late" Video Message and Flyer
Number analyzed (Participants) | 210 | 218 | 202 | 206
score on a scale | 3.710 (2.751) | 3.243 (2.715) | 3.060 (2.509) | 3.685 (2.760)

ADVERSE EVENTS:
Time Frame: Subject participation lasted 15 minutes.
Description: No adverse events were reported.
Arm/Group | "Big Tobacco" Video Message and Flyer | "It's Never Too Late" Video Message and Flyer | Placebo Message | Fear Message Video and Flyer
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/207 | 0/210 | 0/203
Serious Adverse Events (participants affected / at risk) | 0/219 | 0/207 | 0/210 | 0/203
Other Adverse Events (participants affected / at risk) | 0/219 | 0/207 | 0/210 | 0/203

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT05819086/Prot_SAP_000.pdf